CLINICAL TRIAL: NCT00758355
Title: A Prospective, Multicentre Study Evaluating the Clinical Performance of the ReCap/Magnum in Total Hip Replacement and Resurfacing
Brief Title: Data Collection on ReCap/Magnum in Total Hip Replacement and Resurfacing
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Collaborators: Biomet France SARL (Industry)
Responsible Party: Sponsor
Other Study IDs: BMETEU.CR.FR04
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Total Hip Resurfacing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- M2A magnum: Consecutive series of patients received Total Hip Resurfacing with ReCap/Magnum
- Recap Magnum: Consecutive series of patients received Total Hip Replacement with ReCap/Magnum

SUMMARY:
Observational study on ReCap/Magnum in Total Hip Replacement and Resurfacing.

DETAILED DESCRIPTION:
This observational study intends to collect efficacy and safety data on ReCap/Magnum in Total Hip Replacement and Resurfacing.

ELIGIBILITY:
Inclusion Criteria:

Consecutive series of patients received Total Hip Replacement or Resurfacing with ReCap/Magnum for Its Respective Indications for Use/Intended Uses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive series of patients received Total Hip Replacement or Resurfacing with ReCap/Magnum for Their Respective Indications for Use/Intended Uses
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2008-03; Primary Completion 2013-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Postel-Merle d'Aubigné (PMA), Harris Hip Score | 1yr and 2yr

SECONDARY OUTCOMES:
Complication | Any time
Survival | 1yr and 2yr

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Saragaglia, Pr, Principal Investigator — Hopital Sud - Echirolles
Locations (6):
- France (6):
  - CHU Amiens, Amiens
  - CHU Pellegrin Tripode, Bordeaux
  - CHU Hôpital Sud, Grenoble
  - Polyclinique de Hénin Beaumont, Hénin-Beaumont
  - Polyclinique de Riaumont, Liévin
  - Clinique Saint Andre, Reims